CLINICAL TRIAL: NCT03401216
Title: StEnt Coverage and Neointimal Tissue Characterization After eXtra Long evErolimus - Eluting Stent imPlantation: Prospective sTudy Using optIcal cOhereNce Tomography
Brief Title: StEnt Coverage and Neointimal Tissue Characterization After eXtra Long evErolimus - Eluting Stent imPlantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Exeption
Record Dates: First submitted 2017-12-25; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Ischemic Heart Disease; Coronary Artery Disease; Coronary Atherosclerosis
Keywords: Optical coherence tomography; Healing score; Neointimal coverage; synergy 48; long lesion
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: 80 patients, that underwent PCI with Synergy 48 mm stent implantation, will be randomized into 2 groups of follow-up OCT-visualization - 3 and 6 month.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYNERGY 48 PCI + 3 month OCT follow-up (Experimental): Synergy 48 mm stent implantation followed by 3 month OCT imaging
  Interventions: Device: SYNERGY 48 mm; Procedure: PCI; Procedure: 3 month OCT follow-up
- SYNERGY 48 PCI + 6 month OCT follow-up (Experimental): Synergy 48 mm stent implantation followed by 6 month OCT imaging
  Interventions: Device: SYNERGY 48 mm; Procedure: PCI; Procedure: 6 month OCT follow-up

INTERVENTIONS:
Device: SYNERGY 48 mm — Material: Platinum-Chromium alloy. Stent strut thickness: 0.0029-0.0032 inches. Polymer carrier composed of PLGA (poly(DL-lactide-co-glycolide)). Drug product: Everolimus, 1µg per 1 mm2. Stent diameters available: 2.25; 2.50; 2.75; 3.00; 3.50; 4.00 mm. Stent length: 48 mm. Nominal balloon pressure: 11 atm. (1117 kPa). Manufacturing company: Boston Scientific Corporation (USA)
Procedure: PCI — Standard PCI procedure
Procedure: 3 month OCT follow-up — Optical coherence tomography imaging of target vessel within 3 month after PCI
  Arms: SYNERGY 48 PCI + 3 month OCT follow-up
Procedure: 6 month OCT follow-up — Optical coherence tomography imaging of target vessel within 5 month after PCI
  Arms: SYNERGY 48 PCI + 6 month OCT follow-up

SUMMARY:
The objective of this study is to evaluate the rate of SYNERGY 48 mm stent strut coverage and assess neointimal progression via OCT measurement in patients who underwent PCI.

DETAILED DESCRIPTION:
Patients with stable, unstable angina and non-ST-elevation ACS will be included in this study. Patient will undergo coronary angiography for coronary anatomy assessment and estimation indications for PCI . After screening an OCT-guided PCI with extra long SYNERGY stent implantation will be provided in all patients. Patient will be divided into 2 groups of follow-up and will be followed within 3 and 6 month after procedure. Final clinical follow-up will be assessed at 12 month for all patients. At each follow-up visits the data regarding clinical events, coronary angiography and OCT-imaging will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent before study procedures
* Subject is eligible for percutaneous coronary intervention (PCI)
* Left ventricular ejection fraction (LVEF) >30%
* Reference vessel diameter (RVD) ≥2.25 mm and ≤4.0 mm
* Target lesion(s) length must be ≥38 mm
* Target lesion(s) stenosis ≥50%

Exclusion Criteria:

* History of acute or recent stroke (<2 months)
* Contraindications for antiplatelet and/or anticoagulant therapy
* Bleeding within the last 30 days
* Subject has acute ST elevation MI (STEMI)
* Subject has cardiogenic shock, hemodynamic instability requiring inotropic or mechanical circulatory support
* Subject with out of range complete blood count (CBC) values determined as a clinically significant
* Subject has documented or suspected liver disease, including laboratory evidence of hepatitis
* Subject has baseline serum creatinine level >2.0 mg/dL (177µmol/L)
* Subject has signs or symptoms of active heart failure (i.e., NYHA class IV) at the time of the index procedure
* Subject is a woman who is pregnant or nursing (a pregnancy test must be performed within 7 days prior to the index procedure in women of child-bearing potential)
* Lesion located within a saphenous vein graft or an arterial graft
* Subject has unprotected left main coronary artery disease (>50% diameter stenosis)
* Other serious medical illness (e.g., cancer, congestive heart failure) that may reduce life expectancy to less than 12 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-04-30 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Neointimal healing score | within 3 month after PCI
  The neointimal healing score is based on four stent-related characteristics and is calculated on a lesion level:
  * Presence of filling defect (% intraluminal defect, ILD) is assigned a weight of "4".
  * Presence of both malapposed and uncovered struts (% malapposed/ uncovered, MU) is assigned a weight of "3"
  * Presence of uncovered struts alone (% malapposed, M) is assigned a weight of "2"
  * Presence of malapposed struts alone (% uncovered, U) is assigned a weight of "1"
Neointimal healing score | within 6 month after PCI
  The neointimal healing score is based on four stent-related characteristics and is calculated on a lesion level:
  * Presence of filling defect (% intraluminal defect, ILD) is assigned a weight of "4".
  * Presence of both malapposed and uncovered struts (% malapposed/ uncovered, MU) is assigned a weight of "3"
  * Presence of uncovered struts alone (% malapposed, M) is assigned a weight of "2"
  * Presence of malapposed struts alone (% uncovered, U) is assigned a weight of "1"

SECONDARY OUTCOMES:
Percentage of strut coverage assessed by OCT | within 3 month after PCI
  In metallic DES, the struts are classified as covered in the presence of a coverage thickness >0 μm (tissue can be identified above the struts).
Percentage of strut coverage assessed by OCT | within 6 month after PCI
  In metallic DES, the struts are classified as covered in the presence of a coverage thickness >0 μm (tissue can be identified above the struts).
Percentage of mature neointimal tissue assessed by OCT | within 3 month after PCI
  To assess mature neointima an OCT-based grey-scale-signal-intensity (GSI)-analysis will be performed.
Percentage of mature neointimal tissue assessed by OCT | within 6 month after PCI
  To assess mature neointima an OCT-based grey-scale-signal-intensity (GSI)-analysis will be performed.

OTHER OUTCOMES:
Target lesion failure (TLF) | 12 month after PCI
  TLF is defined as a composite endpoint of cardiac death, target vessel myocardial infarction and clinically indicated target lesion revascularization.
Cardiac death | 12 month after PCI
  Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
Myocardial infarction | 12 month after PCI
  Type 1, 2, 3, 4a, 4b according to Third Universal Definition of Myocardial Infarction
Stent thrombosis | 12 month after PCI
  Definite and probable, according to ARC definition,

CONTACTS AND LOCATIONS:
Locations (1):
- Academician E.N. Meshalkin national medical research center, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: Undecided